CLINICAL TRIAL: NCT05976139
Title: Treatment of Macular Oedema in Patients With Hereditary Retinal Dystrophies by Applying the Micropulsed Subthreshold Laser
Brief Title: Micropulsed Laser in Patients With Macular Oedema in Retinal Dystrophies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, lucia ziccardi, Principal Investigator, Fondazione G.B. Bietti, IRCCS
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Neu 01-23
Record Dates: First submitted 2023-07-19; First posted 2023-08-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Macular Edema; Inherited Retinal Dystrophy; Laser Retinopathy
Keywords: Visual Acuity; Retinal Function; IRD; Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- inherited retinal dystrophies with macular oedema (Experimental): Laser treatment will be performed in patients with macular edema in IRD (experimental arm) who:
  * underwent treatment with diuretics or nutritional drainage products for 3 months and subsequent 'wash-out' of one month 17,18 and had no reduction in macular oedema, in terms of central retinal thickness, of at least 20% compared with the initial assessment
  * they have had an intravitreal injection of anti-VEGF or steroids, and after 3 months there is no reduction in central retinal thickness (CRT) of at least 20% compared to the initial assessment
  * have after 3 months a thickness reduction <10% compared to baseline assessment, following initial treatment with micropulsed laser, and may be candidates for repeating treatment;
  * are not eligible for diuretic therapy due to the presence of comorbidities.
  Interventions: Device: subthreshold treatment with micropulsed laser

INTERVENTIONS:
Device: subthreshold treatment with micropulsed laser — The laser instrument used is the Q 577® Laser System, Iridex, wavelength 577 yellow. The standard pattern used is:
  * Power: 5% Duty Cycle
  * Power 250 mw
  * Pulse duration 200 ms
  * Spot size 100 micron
  * Pattern spacing 0.0 confluente, griglie 7x7

SUMMARY:
The purpose of this study is to investigate whether subthreshold treatment with micropulsed laser can be effective in resolving macular edema in patients with inherited retinal dystrophy.

Visits will be performed after 1, 3, 6, 9, 12, 18, and 24 months after treatment. Laser treatment will be performed on the day of the first visit, and its repetition at subsequent visits between months 3 and 12 will be evaluated.

Evaluations of treatment effects will include:

* comprehensive ophthalmologic examination
* multifocal electroretinogram
* OCT examination
* OCT-angiography examination
* retinography

Primary endpoint.

- central retinal thickness, measured by OCT

DETAILED DESCRIPTION:
BACKGROUND:

Degenerative diseases of the visual system classified as rare and, in particular, those affecting the retina (known as Inherited retinal dystrophies, IRDs) cause very severe functional deficits. Their onset is in many cases particularly early with a consequent visual impact of extreme severity. They constitute a heterogeneous group from a clinical point of view, but in all of them the loss of photoreceptors causes progressive vision loss that can result in complete blindness.

These pathologies can be complicated by the presence of cataracts, epiretinal membrane and macular oedema (10-50%), resulting in a worsening of visual acuity. While surgical treatment is applicable for the first two complications, the treatment of macular oedema can make use of several options. Oral or topical diuretics (Acetazolamide) are still the first therapeutic approach and, if oedema persists despite treatment, intravitreal corticosteroid injection has been used in various reports. The injection of anti-Vascular Endothelial Growth Factor (VEGF) drugs and vitrectomy have also been proposed but with conflicting results. The use of topical non-steroidal drugs has been studied and proven to be valuable, although inferior to diuretic treatment in terms of visual recovery. The use of intravitreal corticosteroids is also not without possible further complications such as ocular hypertension and early onset of cataracts.

Despite some improvement in retinal oedema by taking the above-mentioned diuretics, relapses can be observed at the end of therapy, reason for taking longer periods (>12 weeks) of therapy. However, the same chronic continuation of diuretic therapy is not always desirable considering its possible adverse events such as tingling sensation, malaise, altered taste sensation and gastrointestinal disorders.

RATIONALE:

The application of the micropulsed subthreshold retinal laser to reduce retinal oedema in various diseases (diabetic oedema, central serous chorioretinopathy, age-related macular degeneration and retinal vein occlusion) has recently gained wide acceptance.

Retinal threshold refers to the tendency of the laser to cause tissue bleaching resulting in retinal cell death, the term sub-threshold implies that the laser uses such a small amount of energy that it does not cause irreversible damage to retinal structures. The term 'micropulsed' derives from the fact that the laser does not use a continuous wave but has a sub-100% duty cycle and the use of 'off' times is what distinguishes this type of laser from conventional lasers and allows the tissue to cool down, preventing laser-induced retinal damage.

The main characteristics of this type of laser are therefore that it does not cause visible retinal damage and that it has therapeutic effects.

One theory of how this type of laser works is through the action of the molecular protective mechanisms of the Heat Shock Protein (Hsp) family in the retina, including protein chaperone activity, stabilisation of the cytoskeleton and prevention of apoptosis mainly through inhibition of cytochrome C release through the phenomenon of 'resetting'. Another theory hypothesized the activation of leucocyte recruitment or remodeling of the extracellular matrix in the choroid and retina. Possible mechanisms of increased trophic factors (CNTF and FGF-2)14 and up-regulation of other factors (MMP-2, MMP-3, TNFα and Nos2) are covered.

TRIAL DESIGN:

Prospective, interventional, single-centre, open-label study involving consecutive enrolment (see sample size in section "Statistics") of patients with macular oedema in retinal dystrophies.

Each patient referred to the Outpatient Clinical and Research Center of Neuro-ophthalmology and Genetic and Rare Diseases with IRD and macular oedema treated for 3 months with diuretics and draining food supplements and without improvement of macular oedema or increase of the same (reduction of post-therapy CRT ≤20% compared to pre-therapy CRT) will be duly informed about the therapeutic option of this study protocol. After verification of the criteria for inclusion in the study and after signing of the informed consent, the patient will be considered eligible for treatment with micropulsed laser by the physicians of the Clinical and Research Center of Neuro-ophthalmology and Genetic and Rare Diseases and Medical Retina. The patient enrolled in the study will be clinically analysed with the instrumentation indicated below at regular intervals (screening/baseline, follow-up 1 [FU1] (1 month), FU2 (3 months), FU3 (6 months), FU4 (9 months), FU5 (12 months), FU6 (18 months) and FU7 (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with inherited retinal disease
* Age between 18 and 80 years
* Conclusive molecular genetic study for IRD
* Male or female patient
* Presence of macular oedema assessed by sd-OCT with reduction ≤ 20% after 3 months of diuretics or draining supplements or 4 months after last anti-VEGF or steroid injection
* Phakic and pseudophakic patients
* Central Retinal thickness > 320 microns in men and > 305 microns in women
* Informed consent freely granted and acquired before the start of the study
* Participant has the ability to understand and willingness to follow study instructions and is likely to complete all required visits and procedures.

Exclusion Criteria:

* Patients with cataract extraction prior to 6 months
* Patients with IOP ≥ 20 mmHg
* Patients with a clinical diagnosis of retinal dystrophy of unproven genetic origin
* Patients with diabetes
* Patients with central serous chorioretinosis, retinal vein occlusion, age-related degeneration
* Patients with current or previous vitreo-retinal pathology or with indication for vitreo-retinal surgical therapy (tractional oedema)
* Patients with a lack of target fixation at 32 cm
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
assessment of significative change in retinal oedema compared to baseline | up to 24 months
  assessment of central retinal thickness by macular SD-OCT

SECONDARY OUTCOMES:
To study changes in visual acuity between before and after treatment | up to 24 months
  LogMAr visual acuity values
To study the retinal function in the macular area before and after treatment. | up to 24 months
  response amplitude density, measured in nV/dg2 and analysed using multifocal electroretinogram, assessing the amplitude in 5 concentric rings centred on the fovea.
To study the retinal perfusion of the macular area by OCT-angiography before and after treatment. | up to 24 months
  vascular density (expressed as Retinal Vessel Density) before and after treatment, using OCT-angiography

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Ziccardi, MD, PhD, Principal Investigator — IRCCS Fondazione G.B. Bietti
Locations (1):
- IRCSS Fondazione G:B:Bietti, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
At the end of the research, within 6 months after the end of the study, a Final Clinical Report of the study containing clinical comments based on the data generated by the statistical processing will be prepared by the Investigator and/or delegated person. This report will be structured as an "integrated statistical clinical report" containing the clinical comments based on the data generated by the statistical report.
Supporting Information: CSR
Time Frame: Six months after the end of the study
Access Criteria: On demand

REFERENCES:
- [Background] Olivares-Gonzalez L, Velasco S, Campillo I, Rodrigo R. Retinal Inflammation, Cell Death and Inherited Retinal Dystrophies. Int J Mol Sci. 2021 Feb 20;22(4):2096. doi: 10.3390/ijms22042096. PMID 33672611
- [Background] Bakthavatchalam M, Lai FHP, Rong SS, Ng DS, Brelen ME. Treatment of cystoid macular edema secondary to retinitis pigmentosa: a systematic review. Surv Ophthalmol. 2018 May-Jun;63(3):329-339. doi: 10.1016/j.survophthal.2017.09.009. Epub 2017 Oct 5. PMID 28987613
- [Background] Hong Y, Li H, Sun Y, Ji Y. A Review of Complicated Cataract in Retinitis Pigmentosa: Pathogenesis and Cataract Surgery. J Ophthalmol. 2020 Dec 21;2020:6699103. doi: 10.1155/2020/6699103. eCollection 2020. PMID 33489339
- [Background] Ikeda Y, Yoshida N, Murakami Y, Nakatake S, Notomi S, Hisatomi T, Enaida H, Ishibashi T. Long-term Surgical Outcomes of Epiretinal Membrane in Patients with Retinitis Pigmentosa. Sci Rep. 2015 Aug 13;5:13078. doi: 10.1038/srep13078. PMID 26268934
- [Background] Sahel J, Bonnel S, Mrejen S, Paques M. Retinitis pigmentosa and other dystrophies. Dev Ophthalmol. 2010;47:160-167. doi: 10.1159/000320079. Epub 2010 Aug 10. PMID 20703049
- [Background] Lemos Reis RF, Moreira-Goncalves N, Estrela Silva SE, Brandao EM, Falcao-Reis FM. Comparison of topical dorzolamide and ketorolac treatment for cystoid macular edema in retinitis pigmentosa and Usher's syndrome. Ophthalmologica. 2015;233(1):43-50. doi: 10.1159/000368052. Epub 2014 Nov 26. PMID 25428176
- [Background] Orzalesi N, Pierrottet C, Porta A, Aschero M. Long-term treatment of retinitis pigmentosa with acetazolamide. A pilot study. Graefes Arch Clin Exp Ophthalmol. 1993 May;231(5):254-6. doi: 10.1007/BF00919100. PMID 8319913
- [Background] Moore SM, Chao DL. Application of subthreshold laser therapy in retinal diseases: a review. Expert Rev Ophthalmol. 2018;13(6):311-320. doi: 10.1080/17469899.2018.1555035. Epub 2018 Dec 11. PMID 31692951
- [Background] Franklin TB, Krueger-Naug AM, Clarke DB, Arrigo AP, Currie RW. The role of heat shock proteins Hsp70 and Hsp27 in cellular protection of the central nervous system. Int J Hyperthermia. 2005 Aug;21(5):379-92. doi: 10.1080/02656730500069955. PMID 16048836
- [Background] Caballero S, Kent DL, Sengupta N, Li Calzi S, Shaw L, Beli E, Moldovan L, Dominguez JM 2nd, Moorthy RS, Grant MB. Bone Marrow-Derived Cell Recruitment to the Neurosensory Retina and Retinal Pigment Epithelial Cell Layer Following Subthreshold Retinal Phototherapy. Invest Ophthalmol Vis Sci. 2017 Oct 1;58(12):5164-5176. doi: 10.1167/iovs.16-20736. PMID 29049716
- [Background] Chidlow G, Shibeeb O, Plunkett M, Casson RJ, Wood JP. Glial cell and inflammatory responses to retinal laser treatment: comparison of a conventional photocoagulator and a novel, 3-nanosecond pulse laser. Invest Ophthalmol Vis Sci. 2013 Mar 28;54(3):2319-32. doi: 10.1167/iovs.12-11204. PMID 23439603
- [Background] Flaxel C, Bradle J, Acott T, Samples JR. Retinal pigment epithelium produces matrix metalloproteinases after laser treatment. Retina. 2007 Jun;27(5):629-34. doi: 10.1097/01.iae.0000249561.02567.fd. PMID 17558327
- [Background] Chalam KV, Bressler SB, Edwards AR, Berger BB, Bressler NM, Glassman AR, Grover S, Gupta SK, Nielsen JS; Diabetic Retinopathy Clinical Research Network. Retinal thickness in people with diabetes and minimal or no diabetic retinopathy: Heidelberg Spectralis optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Dec 13;53(13):8154-61. doi: 10.1167/iovs.12-10290. PMID 23132803
- [Background] Elman MJ, Bressler NM, Qin H, Beck RW, Ferris FL 3rd, Friedman SM, Glassman AR, Scott IU, Stockdale CR, Sun JK; Diabetic Retinopathy Clinical Research Network. Expanded 2-year follow-up of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):609-14. doi: 10.1016/j.ophtha.2010.12.033. PMID 21459214
- [Background] Marashi A, Zazo A. Hybrid threshold laser to treat diabetic macular edema: A retrospective analysis single center cohort study. Ann Med Surg (Lond). 2022 Jul 31;80:104222. doi: 10.1016/j.amsu.2022.104222. eCollection 2022 Aug. PMID 36045820
- See also: Hereditary Retinal Degenerations and Cystoid Macular Edema — https://pubmed.ncbi.nlm.nih.gov/27913439/
- See also: Photothermal Stimulation with a Micropulse Laser — https://pubmed.ncbi.nlm.nih.gov/26697211/
- See also: Retinal Distrophies — https://www.ncbi.nlm.nih.gov/books/NBK564379/